CLINICAL TRIAL: NCT02668536
Title: Assessing the Safety and Efficacy of Multifunctional Skin-adhesive Nanoparticles for UV Protection in Humans
Brief Title: A Sunscreen Based on Bioadhesive Nanoparticles
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1512016909
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Melanoma; UV Ray Skin Damage
Keywords: sunscreen; melanoma; improved protection from uv rays
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- UV Filter + BNP (Experimental): A UV filtering agent and bioadhesive nanoparticles (BNPs) will comprise the experimental condition in this study. Participants will have 5 sites on their torso where they will have these placed.
  Interventions: Drug: Standard Sunscreen; Device: BNP
- BNP only (Sham Comparator): A placebo bioadhesive nanoparticles (BNPs) (strips with no UV filtering) will comprise the sham comparison in this study. Participants will have 5 sites on their torso where they will have these placed.
  Interventions: Device: BNP
- Standard (Active Comparator): As the active comparator, participants will have 5 sites on their torso where they will have standard sunscreen applied.
  Interventions: Drug: Standard Sunscreen
- Control (No Intervention): Participants will have 5 sites on their torso where no agent will be applied.

INTERVENTIONS:
Drug: Standard Sunscreen — Areas will be treated with a standard preparation, consisting of padimate O (7%) and oxybenzone (3%) will be used as the control sunscreen.
  Arms: Standard; UV Filter + BNP
Device: BNP — Additional areas will be treated with empty bioadhesive nanoparticles (BNPs).
  Arms: BNP only; UV Filter + BNP

SUMMARY:
The initial focus of the study will be on safety, sun protection factor (SPF) characterization, and substantivity (duration of protection) studies. The primary outcome of the study will be to measure the sun protection factor (SPF) of a bioadhesive nanoparticles (BNP) formulation in 20-25 healthy volunteers with fair skin.

DETAILED DESCRIPTION:
The purpose of this study will be to evaluate the duration of protection and efficacy of a novel bioadhesive nanoparticle sunscreen in 20-25 human volunteers.This technology makes sunscreens safer and longer-lasting by encapsulating UV sunscreen active agents in non-toxic nanoparticles. Strong preclinical data exists demonstrating the potential for improved safety, long-duration of retention, and increased effectiveness of this product.

This innovative solution focuses on preventing damage caused by UV exposure through the use of a nanoparticle delivery vehicle. The bioadhesive feature of this technology enables longer protection. In addition, encapsulation of the UV filter in a bioadhesive nanoparticle (BNP) improves filter photo-stability, delays filter photo-degradation, and prevents reactive oxygen species (ROS) escape, thereby reducing the risk of cell damage and epidermal toxicity from UV filters.

Furthermore, the bioadhesive feature of our technology eliminates penetration into deeper skin layers or into the blood, minimizing the potential side-effects of UV filters. It is believed that the translation of this technology will provide a longer-lasting, safer, more protective UV sunscreen.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be in good health with minimal skin irregularities, as evaluated by a physical examination.
* The physical examination shall determine the presence of sunburn, suntan, scars, active dermal lesions, and uneven skin tones on the areas of the back to be tested. The presence of nevi, blemishes, or moles will be acceptable if in the physician's judgment they will not interfere with the study results. Excess hair on the back is acceptable if the hair is clipped or shaved.
* Subjects must fall into one of the following 3 Fitzpatrick Skin Scale categories:

  1. Always burns easily; never tans (sensitive)
  2. Always burns easily; tans minimally (sensitive)
  3. Burns moderately; tans gradually (light brown) (normal)

Exclusion Criteria:

* Volunteers cannot have a history of skin cancer (such as basal cell carcinoma, squamous cell carcinoma, or melanoma).
* Volunteers cannot have a history of skin disease (such as psoriasis, exema, or vitiligo).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-18 (Actual)

PRIMARY OUTCOMES:
Skin Reaction | 1 week
  Skin reaction will be assessed by exam. The exam will look for evidence of irritation, inflammation, follicular occlusion. In addition, patients will report any skin reaction at site of application over one week. Severity of the skin reactions will be assessed in the following manner: severe reactions will include evidence of edema or blister formation, follicular pustules and/or marked erythema and pruritus.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Girardi, MD, FAAD, Principal Investigator — Yale University; Mark Saltzman, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No